CLINICAL TRIAL: NCT04961840
Title: Observational Study to Assess Maternal and Fetal Outcomes Following Exposure to Prucalopride During Pregnancy
Brief Title: A Study to Assess Maternal and Fetal Outcomes After Taking Prucalopride During Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-555-5002; EUPAS41866 (Other: EUPAS Register Number)
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Constipation; Pregnancy
Keywords: Prucalopride; infant outcomes
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Pregnant Women Exposed to Prucalopride: Pregnant women with clinically diagnosis of constipation who have been exposed to prucalopride during pregnancy will be observed.
  Interventions: Other: No Intervention
- Cohort 2: Pregnant Women Not Exposed to Prucalopride: Pregnant women with clinical diagnosis of constipation who have been exposed to other constipation drugs and not prucalopride during pregnancy will be observed.
  Interventions: Other: No Intervention
- Cohort 3: Untreated Pregnant Women: Pregnant women with clinical diagnosis of constipation with no recorded prescription dispensed for any constipation drugs during pregnancy will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This study will collect information on pregnant women diagnosed with constipation from the two large health care insurance claims records.

It will include the following groups:

* Those who took prucalopride.
* Those who took other medicines for constipation.
* Those who did not take any prescription medicines for constipation.

The main aim of the study is to find out whether the medicine prucalopride, which is used to treat constipation, is safe for use during pregnancy and to look at whether taking prucalopride at certain times during pregnancy is associated to a higher chance of specific health problems for the mother or baby.

The study uses two large existing healthcare insurance databases for collecting information. Participants are not enrolled, treated, or required to visit the doctor during this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 to 44 years with constipation.
* Maternal coverage by health care and prescriptions insurance during eligibility period:

  a) To study pregnancy outcomes (live births, spontaneous abortions, terminations, or stillbirths): 90 days prior to the LMP until end of pregnancy; and b) to study malformations, perinatal and infant outcomes: 90 days to LMP until 30 days post-delivery.
* For infant outcomes, the cohort will be restricted to pregnancies with linked offspring.
* For major malformations, only pregnancies with livebirths will be included, since information regarding the pathological results from a pregnancy loss or the indication for termination is rarely recorded. In addition, infants are required to have full insurance coverage from delivery to at least 90 days after the delivery, unless the infant died prior to the end of the 90 days, in which case a shorter eligibility period until death is permitted.
* For the analyses of pregnancy losses, the cohort also includes pregnancies ending in spontaneous abortion, terminations, stillbirth and any livebirth (linked or unlinked to a delivery).

Exclusion Criteria:

* Women with opioids dispensed in the 3 months prior to LMP or during the first trimester (to exclude potential opioid-induced constipation) and women with inflammatory bowel diseases (IBD) (because IBD is a contraindication)
* For major malformations, the cohort excludes pregnancies with a chromosomal abnormality based on at least one inpatient or outpatient ICD-9 code for 758.xx,759.81-759.83, or 655.1x within 90 days after delivery in the infant and/or maternal claims.
* For major malformations, pregnancies with outpatient exposure to definite teratogens including warfarin, valproate, antineoplastic agents, colchicine, testosterone, radioiodine, isotretinoin, misoprostol, and thalidomide from LMP through LMP plus 90 days.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Study Population: This study will include pregnancy women with constipation including those with constipation predominant irritable bowel syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Infants With Major Congenital Malformations | From delivery up to 90 days post-delivery
  A major congenital malformation is defined as a structural abnormality with surgical, medical, or cosmetic importance. Major malformations will be sorted and grouped according to the International Classification of Diseases 10th Revision (ICD-10). Percentage of infants with major congenital malformations after birth will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With Spontaneous Abortions | 90 days prior to the Last menstrual period (LMP) until end of pregnancy
  Spontaneous abortions will be defined as spontaneous losses before 20 weeks of gestation. Percentage of participants with spontaneous abortion will be reported.
Percentage of Participants With Terminations (Discontinuation of Pregnancy) | 90 days prior to the LMP until end of pregnancy
  Percentage of participants with discontinuation of pregnancy through medication or surgical procedures will be reported.
Percentage of Participants With Stillbirths | 90 days prior to the LMP until end of pregnancy
  Stillbirths will be defined as in utero fetal deaths at or after 20 weeks of gestation. Percentage of participants with stillbirths will be reported.
Percentage of Participants With Preterm Delivery | From Delivery to 30 days post-delivery
  Preterm delivery is defined as a live birth occurring at less than (<) 37 gestational weeks.
Percentage of Infants With Small for Gestational Age (SGA) | From Delivery to 30 days post-delivery
  SGA will be defined as weight at birth of full and preterm live-born infants in <10th percentile. Percentage of infants with SGA will be reported.
Percentage of Infants With Neonatal Intensive Care Unit (NICU) Admission | From Delivery to 30 days post-delivery
  Percentage of infants admitted to NICU in relation to early and late pregnancy. exposure to prucalopride will be reported.
Percentage of Infants With Hospitalizations | From Delivery to 365 days post-delivery
  Percentage of infants With Hospitalizations during the first year of life in relation to prenatal exposure to prucalopride will be reported.
Percentage of Infants With Poor Growth and Developmental Delays or Disorders | From Delivery to 365 days post-delivery
  Percentage of infants With Poor Growth and developmental delays or disorders during the first year of life in relation to prenatal exposure to prucalopride will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60f18511268b2a001f5a991f